CLINICAL TRIAL: NCT00621075
Title: Correlation of Hemodynamics in Pulmonary Hypertension With Perfusion Lung Scans
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: ARUNABH TALWAR MD, NORTH SHORE-LONG ISLAND JEWIAH HEALTH SYSTEM
Other Study IDs: 07.014; NORTH SHORE IRB
Record Dates: First submitted 2008-01-17; First posted 2008-02-22 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; V/Q SCAN;RHC;Echo;CT Scans; Angiography;PFTs
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — hydralazine 4-anisaldehyde hydrazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Pulmonary Arterial Hypertension
  Interventions: Other: Pulmonary Arterial Hypertension - Lung Perfusion Scans

INTERVENTIONS:
Other: Pulmonary Arterial Hypertension - Lung Perfusion Scans — Correlation of data from non-invasive tests such as lung perfusion scans with hemodynamic measurements
  Other Names: Pulmonary Arterial Hypertension

SUMMARY:
The goal of our study is to correlate data from non-invasive tests such as perfusion lung scans with hemodynamic measurements from right heart catherizations.

DETAILED DESCRIPTION:
Data collected from PAH patients who have had non-invasive Ventilation/Perfusion testing, Echocardiography, Chest CT Scan, Pulmonary Function Testing and the correlation of those results to the hemodynamic parameters Right Heart Catherization results and the various biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary Arterial Hypertension

Exclusion Criteria:

* Non-Pulmonary Arterial Hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonary Arterial Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The correlation of patients' hemodynamic parameters with their perfusion index/pulmonary index as measured by ventilation perfusion scans in patients diagnosed with Pulmonary Hypertension. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: ARUNABH TALWAR, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore-Lij Health System, New Hyde Park, New York, United States